CLINICAL TRIAL: NCT01449929
Title: A Phase IIIb, Randomized, Open-label Study of the Safety and Efficacy of GSK1349572 (Dolutegravir, DTG) 50 mg Once Daily Compared to Darunavir/Ritonavir (DRV/r) 800 mg/100 mg Once Daily Each Administered With Fixed-dose Dual Nucleoside Reverse Transcriptase Inhibitor Therapy Over 96 Weeks in HIV-1 Infected Antiretroviral naïve Adult Subjects
Brief Title: Dolutegravir Compared to Darunavir/Ritonavir , Each in Combination With Dual Nucleoside Reverse Transcriptase Inhibitors (NRTIs) in ART-naive Subjects
Acronym: FLAMINGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114915
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2014-03-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-10

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: ritonavir; HIV; HAART; darunavir; antiretroviral; dolutegravir; GSK1349572
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- dolutegravir 50mg once daily (OAD) (Experimental): in combination with either abacavir/lamivudine fixed dose combination tablet OAD or tenofovir disoproxil fumarate/emtricitabline fixed dose combination tablet OAD
  Interventions: Drug: dolutegravir 50 mg OAD
- darunavir 800mg OAD in combination with ritonavir 100mg OAD (Active Comparator): in combination with either abacavir/lamivudine fixed dose combination tablet OAD or tenofovir disoproxil fumarate/emtricitabline fixed dose combination tablet OAD
  Interventions: Drug: darunavir 800mg OAD; Drug: ritonavir 100mg OAD

INTERVENTIONS:
Drug: dolutegravir 50 mg OAD — 1 x 50 mg tablet OAD
  Arms: dolutegravir 50mg once daily (OAD)
Drug: darunavir 800mg OAD — 2 x 400mg tablets OAD
  Arms: darunavir 800mg OAD in combination with ritonavir 100mg OAD
Drug: ritonavir 100mg OAD — 1 x 100mg tablet OAD
  Arms: darunavir 800mg OAD in combination with ritonavir 100mg OAD

SUMMARY:
This study will be conducted in approximately 468 HIV-1 infected antiretroviral therapy (ART)-naïve subjects. Subjects will be randomized 1:1 to receive dolutegravir (DTG) 50 mg once daily (approximately 234 subjects) or darunavir/ritonavir (DRV/r) 800 mg/100 mg once daily (approximately 234 subjects), each in combination with fixed-dose dual nucleoside reverse transriptase inhibitor (NRTI) therapy (either abacavir/lamivudine (ABC/3TC) or tenofovir/emtricitabine (TDF/FTC). Subjects will be stratified by screening HIV-1 RNA and background NRTI selection. The primary analysis will take place after the last subject completes 48 weeks on therapy; an additional analysis will be conducted after the last subject completes Week 96 on study.

DETAILED DESCRIPTION:
ING114915 is a Phase IIIb randomized, open-label, active-controlled, multicentre, parallel group, fully-powered non-inferiority study. The study will be conducted in approximately 468 HIV-1 infected ART-naïve subjects. Subjects will be randomized 1:1 to receive DTG 50 mg once daily (approximately 234 subjects) or DRV/r 800 mg/100 mg once daily (approximately 234 subjects), each in combination with fixed-dose dual NRTI therapy (either ABC/3TC or TDF/FTC). The primary analysis will take place after the last subject completes 48 weeks on therapy; an additional analysis will be conducted after the last subject completes Week 96 on study.

Subjects who fulfil eligibility requirements will be randomized 1:1 to receive DTG 50 mg once daily or DRV/r 800 mg/100 mg once daily. In order to achieve balance across the two treatment groups of the study, randomization will be stratified by: screening plasma HIV-1 RNA >/ 100,000 copies/mL (c/mL) or > 100,000 c/mL and background dual NRTI (ABC/3TC or TDF/FTC) The DTG and DRV/r doses will be administered in an open-label fashion throughout the study.

Subjects randomized to receive DTG and who successfully complete 96 weeks of treatment will continue to have access to DTG until either it is locally approved and commercially available, the patient no longer derives clinical benefit, the patient meets a protocol-defined reason for discontinuation or until development of DTG is terminated. Subjects randomized to the DRV/r arm will receive DRV/r through their Week 96 visit, after which they will be discontinued from the study and will need to make alternative arrangements to access antiretroviral medication. All subjects will receive background dual-NRTI therapy through their Week 96 visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults greater than or equal to 18 years of age. Females are eligible to enter and participate in the study if she is (1) non-childbearing potential, (2) child bearing potential with negative pregnancy test at screening and Day 1 and agrees to use protocol-specified methods of birth control while on study.
* HIV-1 infection with a screening plasma HIV-1 RNA greater than or equal to 1000copies/mL
* Antiretroviral-naïve (less than or equal to 10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection)
* Signed and dated written informed consent is obtained from the subject or the subject's legal representative prior to screening

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any evidence of an active Centers for Disease and Prevention Control (CDC) Category C disease [CDC, 1993], except cutaneous Kaposi's sarcoma not requiring systemic therapy
* Subjects with moderate to severe hepatic impairment (Class B or C) as determined by Child-Pugh classification
* Anticipated need for Hepatitis C virus (HCV) therapy during the study
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening: radiation therapy; cytotoxic chemotherapeutic agents; any immunomodulators
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 in vitro within 28 days of first dose of investigational product
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of investigational product
* Any evidence of primary viral resistance based on the presence of any major resistance-associated mutation [IAS-USA, 2010] in the Screening result or, if known, any historical resistance test result
* Any verified Grade 4 laboratory abnormality. Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound is exclusionary
* Alanine aminotransferase (ALT) greater than 5 times the upper limit of normal
* ALT greater than 3 times the upper limit of normal and bilirubin greater than or equal to 1.5 times the upper limit of normal (with greater than 35% direct bilirubin)
* Subject has creatinine clearance of less than 50 mL/min via Cockroft-Gault method
* Recent history (less than or equal to 3 months) of any upper or lower gastrointestinal bleed, with the exception of anal or rectal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2013-04-22 (Actual); Study Completion 2016-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (55):
- United States (28):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Seattle, Washington
- France (4):
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Denis
- Germany (3):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hamburg
- Italy (4):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
- Russia (5):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Volgograd
- Spain (4):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- Switzerland (3):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Zurich

REFERENCES:
- [Derived] Molina JM, Clotet B, van Lunzen J, Lazzarin A, Cavassini M, Henry K, Kulagin V, Givens N, de Oliveira CF, Brennan C; FLAMINGO study team. Once-daily dolutegravir versus darunavir plus ritonavir for treatment-naive adults with HIV-1 infection (FLAMINGO): 96 week results from a randomised, open-label, phase 3b study. Lancet HIV. 2015 Apr;2(4):e127-36. doi: 10.1016/S2352-3018(15)00027-2. Epub 2015 Mar 10. PMID 26424673
- [Derived] Clotet B, Feinberg J, van Lunzen J, Khuong-Josses MA, Antinori A, Dumitru I, Pokrovskiy V, Fehr J, Ortiz R, Saag M, Harris J, Brennan C, Fujiwara T, Min S; ING114915 Study Team. Once-daily dolutegravir versus darunavir plus ritonavir in antiretroviral-naive adults with HIV-1 infection (FLAMINGO): 48 week results from the randomised open-label phase 3b study. Lancet. 2014 Jun 28;383(9936):2222-31. doi: 10.1016/S0140-6736(14)60084-2. Epub 2014 Apr 1. PMID 24698485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2 sequential treatment period study. In first period (Randomization phase) participants received either dolutegravir (DTG) 50 milligram (mg) or darunavir (DRV) 800 mg with ritonavir (RTV) 100 mg once daily (QD) for 96 weeks. DTG participants who completed 96 Weeks of DTG then continued to receive DTG 50 mg in Extension phase.
Pre-assignment Details: A total of 595 participants were screened; 107 were screen failures; 488 were randomized; 485 received at least 1 dose of study medication and comprised the Intent-To-Treat exposed (ITT-E) population of which 1 participant was removed, creating the modified ITT-E population with 484 participants. 123 participants enrolled in Extension Phase.
Groups:
- DTG 50 mg QD: Participants received DTG 50 mg QD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks. Participants were then given the opportunity to receive DTG 50 mg QD during an Extension Phase of the study.
- DRV 800 mg + RTV 100 mg QD: Participants received DRV 800 mg + RTV 100 mg QD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks.
- Extension DTG 50 mg: DTG participants who successfully completed 96 Weeks of randomized phase continued to receive DTG 50 mg QD during Extension phase
Period: Randomization Phase 96 Week
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD | Extension DTG 50 mg
Started | 242 | 242 | 0
Completed | 209 | 189 | 0
Not Completed | 33 | 53 | 0
Not completed — Adverse Event | 5 | 13 | 0
Not completed — Lack of Efficacy | 3 | 4 | 0
Not completed — Protocol Violation | 5 | 6 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 0
Not completed — Lost to Follow-up | 15 | 18 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0
Not completed — Physician Decision | 2 | 3 | 0
Not completed — Other: study closed/terminated | 0 | 1 | 0
Period: Extension Phase Approximately 3 Years
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD | Extension DTG 50 mg
Started | 0 | 0 | 123
Completed | 0 | 0 | 115
Not Completed | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD | Total
Number analyzed (Participants) | 242 | 242 | 484
Age, Continuous [Mean (Standard Deviation); unit: Years] — Results from the mITT-E Population are presented in this report.
  Years | 35.7 (10.66) | 36.2 (10.64) | 35.9 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Results from the mITT-E are presented in this report.
  Participants
    Female | 31 | 41 | 72
    Male | 211 | 201 | 412
Race/Ethnicity, Customized [Number; unit: Participants] — Results from the mITT-E are presented in this report.
  Participants
    African American/African Heritage | 60 | 53 | 113
    American Indian or Alaska Native | 3 | 9 | 12
    Asian - Central/South Asian Heritage | 0 | 1 | 1
    Asian - Japanese Heritage | 1 | 0 | 1
    Asian - South East Asian Heritage | 1 | 0 | 1
    Native Hawaiian or other Pacific Islander | 2 | 0 | 2
    White - Arabic/North African Heritage | 4 | 3 | 7
    White - White/Caucasian/European Heritage | 169 | 173 | 342
    Mixed Race | 1 | 3 | 4
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/Milliliter (c/mL) at Week 48
Description: Assessment was done using Missing, Switch or Discontinuation = Failure (MSDF), as codified by the Food and Drug Administration (FDA) "snapshot" algorithm.This algorithm treated all participants without HIV-1 RNA data at Week 48 as nonresponders, as well as participants who switched their concomitant ART prior to Week 48 as follows: background ART substitutions non-permitted per protocol (one background ART substitution was permitted for safety or tolerability); background ART substitutions permitted per protocol unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment in the snapshot window (Week 48 +/- 6 weeks). Modified Intent-To-Treat Exposed (mITT-E) Population:all randomized participants who received at least one dose of investigational product
Time Frame: Week 48
Population: mITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Percentage of participants | 90 | 83
Statistical Analysis 1: Comparison: DTG 50 mg QD vs DRV 800 mg + RTV 100 mg QD; Test type: Non-Inferiority or Equivalence — Non-inferiority of DTG 50 mg and DRV+RTV at Week 48 can be concluded if the lower bound of a two-sided 95% confidence interval (CI) for the difference in percentages (DTG - DRV+RTV) is greater than -12%. If non-inferiority is established, superiority can be tested at the nominal 5% level based on a pre-specified testing procedure; p = 0.025, Cochran-Mantel-Haenszel — P-value is for test of superiority; Stratified analysis; Difference in percentage = 7.1, 95% CI 2-sided [0.9 to 13.2] — Analysis was adjusted for the Baseline (BL) stratification factors: Baseline plasma HIV-1 RNA (<=100,000 c/mL vs >100,000 c/mL) and Baseline background dual NRTI therapy (ABC/3TC vs TDF/FTC)

2. Secondary Outcome: Time to Virologic Suppression (<50 Copies/mL) Through Week 48
Description: The time to viral suppression (i.e. first viral load value <50 copies/mL) through Week 48 was derived and summarized using Kaplan-Meier plots. Participants who withdrew for any reason without having suppressed prior to the analysis were censored. Confidence intervals were estimated using the Brookmeyer-Crowley method.
Time Frame: From Baseline through Week 48
Population: mITT-E Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Days | 28.0 [NA to NA] — The DTG median time to suppression 95% CI was not estimable due to the steep increase in cumulative incidence at Day 28, so the confidence limit lines do not extend to cross the median line. | 85.0 [84.0 to 108.0]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <400 c/mL at Week 48
Description: The percentage of participants with Plasma HIV-1 RNA <400 c/mL at Week 48 was assessed MSDF, as codified by the FDA "snapshot" algorithm. This algorithm treated all participants without HIV-1 RNA data at Week 48 as nonresponders, as well as participants who switched their concomitant ART prior to Week 48 as follows: background ART substitutions non-permitted per protocol (one background ART substitution was permitted for safety or tolerability); background ART substitutions permitted per protocol unless the decision to switch was documented as being before or at the first on-treatment visit where HIV-1 RNA was assessed. Otherwise, virologic success or failure was determined by the last available HIV-1 RNA assessment while the participant was on-treatment in the snapshot window (Week 48 +/- 6 weeks).
Time Frame: Week 48
Population: mITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Percentage of participants | 92 | 87

4. Secondary Outcome: Change From Baseline in Plasma HIV-1 RNA (log10 c/mL) at Weeks 4, 8, 12, 16, 24, 36 and 48
Description: Change from Baseline in plasma HIV-1 RNA (log10 c/mL) was assessed at Weeks 4, 8, 12, 16, 24, 36 and 48 . Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits, so the overall number of participants analyzed reflects everyone in the mITT-E Population.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 24, 36 and 48
Population: mITT-E Population.
Measure: Mean (Standard Deviation); unit: Log10 copies per mL
Groups:
- DTG 50 mg OD: Participants received DTG 50 mg OD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks. Participants were then given the opportunity to receive DTG 50 mg OD during an Extension Phase of the study.
- DRV 800 mg + RTV 100 mg OD: Participants received DRV 800 mg + RTV 100 mg OD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks.
Arm/Group | DTG 50 mg OD | DRV 800 mg + RTV 100 mg OD
Number analyzed (Participants) | 242 | 242
Log10 copies per mL
  Week 4, n=238, 235: number analyzed (Participants) | 238 | 235
  Week 4, n=238, 235 | -2.80 (0.625) | -2.01 (0.454)
  Week 8, n=237, 236: number analyzed (Participants) | 237 | 236
  Week 8, n=237, 236 | -2.86 (0.649) | -2.40 (0.524)
  Week 12, n=234, 227: number analyzed (Participants) | 234 | 227
  Week 12, n=234, 227 | -2.88 (0.653) | -2.61 (0.537)
  Week 16, n=229, 228: number analyzed (Participants) | 229 | 228
  Week 16, n=229, 228 | -2.86 (0.691) | -2.71 (0.618)
  Week 24, n=234, 227: number analyzed (Participants) | 234 | 227
  Week 24, n=234, 227 | -2.86 (0.765) | -2.83 (0.663)
  Week 36, n=232, 218: number analyzed (Participants) | 232 | 218
  Week 36, n=232, 218 | -2.87 (0.715) | -2.85 (0.683)
  Week 48, n=227, 212: number analyzed (Participants) | 227 | 212
  Week 48, n=227, 212 | -2.89 (0.739) | -2.86 (0.663)

5. Secondary Outcome: Change From Baseline in CD4+ and CD8+ Cell Counts
Description: Change from Baseline in CD4+ cell counts was assessed at Weeks 4, 8, 12, 16, 36 and 48. Change from Baseline in CD8+ cell counts was assessed at Weeks 4, 12, 24 and 48. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits and parameters, so the overall number of participants analyzed reflects everyone in the mITT-E Population.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 36 and 48 for CD4+ and Baseline and Weeks 4, 12, 24 and 48 for CD8+
Population: mITT-E Population.
Measure: Mean (Standard Deviation); unit: Cells per millimeters cubed (cells/mm^3)
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Cells per millimeters cubed (cells/mm^3)
  CD4+ cell count, Week 4, n=237, 236: number analyzed (Participants) | 237 | 236
  CD4+ cell count, Week 4, n=237, 236 | 80.1 (101.36) | 75.6 (124.36)
  CD4+ cell count, Week 8, n=236, 236: number analyzed (Participants) | 236 | 236
  CD4+ cell count, Week 8, n=236, 236 | 126.9 (124.13) | 118.8 (142.54)
  CD4+ cell count, Week 12, n=234, 228: number analyzed (Participants) | 234 | 228
  CD4+ cell count, Week 12, n=234, 228 | 135.2 (120.03) | 131.8 (143.88)
  CD4+ cell count, Week 16, n=227, 227: number analyzed (Participants) | 227 | 227
  CD4+ cell count, Week 16, n=227, 227 | 156.8 (146.60) | 146.1 (166.08)
  CD4+ cell count, Week 24, n=233, 227: number analyzed (Participants) | 233 | 227
  CD4+ cell count, Week 24, n=233, 227 | 165.1 (145.85) | 164.3 (180.00)
  CD4+ cell count, Week 36, n=232, 218: number analyzed (Participants) | 232 | 218
  CD4+ cell count, Week 36, n=232, 218 | 206.1 (159.06) | 186.5 (183.61)
  CD4+ cell count, Week 48, n=227, 212: number analyzed (Participants) | 227 | 212
  CD4+ cell count, Week 48, n=227, 212 | 243.8 (180.68) | 215.4 (177.26)
  CD8+ cell count, Week 4, n=235, 235: number analyzed (Participants) | 235 | 235
  CD8+ cell count, Week 4, n=235, 235 | -47.4 (276.01) | -3.7 (375.94)
  CD8+ cell count, Week 12, n=231, 227: number analyzed (Participants) | 231 | 227
  CD8+ cell count, Week 12, n=231, 227 | -42.0 (343.81) | -68.9 (373.38)
  CD8+ cell count, Week 24, n=231, 224: number analyzed (Participants) | 231 | 224
  CD8+ cell count, Week 24, n=231, 224 | -108.0 (350.03) | -132.9 (389.70)
  CD8+ cell count, Week 48, n=224, 210: number analyzed (Participants) | 224 | 210
  CD8+ cell count, Week 48, n=224, 210 | -109.5 (360.94) | -162.1 (421.07)

6. Secondary Outcome: Number of Participants With HIV-1 Associated Disease Progression With the Indicated Shift to CDC Class C, or New CDC Class C or Death at Week 48
Description: The number of participants with HIV-1 disease progression (AIDS or death) was assessed per the Centers for Disease Control and Prevention (CDC) 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: Week 48
Population: mITT-E Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Participants | 0 | 0

7. Secondary Outcome: Change From Baseline in Fasting Low-density Lipoprotein (LDL) Cholesterol Through Week 48
Description: Fasting LDL cholesterol change from Baseline was analyzed. Values represented are for adjusted means. Estimates are calculated from a repeated measures model including the following covariates: treatment, visit, Baseline plasma HIV-1 RNA, background dual NRTI therapy, Baseline LDL cholesterol, treatment*visit interaction and Baseline LDL cholesterol*visit interaction. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants with data available at the specified time points were analyzed.
Time Frame: From Baseline through Week 48
Population: mSafety Population.
Measure: Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 182 | 178
Millimoles per liter (mmol/L) | 0.07 (0.041) | 0.37 (0.041)

8. Secondary Outcome: Percentage of Participants With Grade 2 or Higher Abnormalities in Fasting LDL Cholesterol Through Week 48
Description: Hematology and clinical chemistry data were summarized according to the division of AIDS (DAIDS) table for grading the Severity of adverse events, version 1.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for which an increase in fasting LDL cholesterol to Grade 2 or higher occurred. Only those participants with data available at the specified time points were analyzed.
Time Frame: From Baseline through Week 48
Population: mSafety Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Percentage of Participants | 2 | 7

9. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Maximum Post-Baseline Chemistry and Hematology Laboratory Toxicities
Description: Hematology and clinical chemistry data were summarized according to the division of AIDS (DAIDS) table for grading the Severity of adverse events, version 1.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred.
Time Frame: From Baseline through Week 48
Population: mSafety Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Participants
  Alanine Amino Transferase, G3 | 2 | 1
  Alanine Amino Transferase, G4 | 1 | 3
  Aspartate Amino Transferase, G3 | 6 | 3
  Aspartate Amino Transferase, G4 | 2 | 0
  Cholesterol, G3 | 0 | 3
  Creatine Kinase, G3 | 8 | 5
  Creatine Kinase, G4 | 8 | 4
  Hyperglycaemia, G3 | 1 | 2
  Hypoglycaemia, G3 | 0 | 1
  LDL Cholesterol, G3 | 2 | 6
  Lipase, G3 | 5 | 5
  Lipase, G4 | 2 | 0
  Phosphorus, inorganic, G3 | 7 | 7
  Total Bilirubin, G3 | 1 | 0
  Triglycerides, G3 | 1 | 2
  Triglycerides, G4 | 0 | 1
  Hemoglobin, G3 | 1 | 0
  Hemoglobin, G4 | 1 | 0
  Platelet count, G4 | 0 | 1
  Total Neutrophils, G3 | 5 | 0
  Total Neutrophils, G4 | 3 | 1

10. Secondary Outcome: Number of Participants (Par.) With Detectable Virus That Has Genotypic or Phenotypic Evidence of Treatment-emergent Resistance to DTG, DRV+RTV and Other On-study ART at Time of Protocol Defined Virology Failure (PDVF)
Description: An assessment was made of every change across all amino acids within the integrase (IN), reverse transcriptase (RT), and Protease (PRO) encoding region at Baseline and at time of suspected PDVF. PDVF is defined as the confirmed plasma HIV-1 RNA >200 c/mL >=Week 24. PDVF Genotypic Population included all participants in the mITT-E population with available on-treatment genotypic resistance data, at time of PDVF. Only those participants with data available at the specified time points were analyzed.
Time Frame: Baseline until PDVF up to Week 48
Population: PDVF Genotypic Population
Measure: Number; unit: Participants
Arm/Group | DTG 50 mg OD | DRV 800 mg + RTV 100 mg OD
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

11. Secondary Outcome: Change From Baseline in Acquired Immune Deficiency Syndrome (AIDS) Clinical Trials Group (ACTG) Symptom Distress Module (SDM) Bother Score at Week 4, Week 24, and Week 48
Description: SDM is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Each item is rated from 0 to 4 where 0 (complete absence of symptom) and 4 (very bothersome symptom). Overall score calculated as the sum of the scores for each of the 20 items of the questionnaire and ranged from 0 (best health) and 80 (worst health). Values represented are for adjusted mean. Estimates are calculated from an ANCOVA model adjusting for age, sex, race, baseline viral load, background dual NRTI therapy and baseline symptom bother score. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. A positive change from Baseline indicates a decline in a participant's quality of life over that period.
Time Frame: Baseline, Week 4, Week 24, and Week 48
Population: mITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits, so the overall number of participants analyzed reflects everyone in the mITT-E Population.
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- DRV 800 mg + RTV 100 mg QD: Participants received DRV 800 mg + RTV 100 mg OD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks.
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Scores on a scale
  Week 4, n=218, 210: number analyzed (Participants) | 218 | 210
  Week 4, n=218, 210 | -3.20 (0.56) | -2.19 (0.56)
  Week 24, n=222, 214: number analyzed (Participants) | 222 | 214
  Week 24, n=222, 214 | -2.71 (0.64) | -1.65 (0.65)
  Week 48, n= 222, 215: number analyzed (Participants) | 222 | 215
  Week 48, n= 222, 215 | -2.46 (0.68) | -0.77 (0.69)

12. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimensions (EQ-5D) Utility Scores at Week 24 and Week 48
Description: The EQ-5D is a 5-question quality of life instrument that provides a utility score and visual analogue scale score that describes the participants' health status. The primary reason for including the EQ-5D is to elicit utility values for potential cost-effectiveness analysis for submission to health technology assessment agencies. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome. Values represented are for adjusted mean. Estimates are calculated from an ANCOVA model adjusting for age, sex, race, baseline viral load, background dual NRTI therapy and Baseline EQ-5D utility score. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24, and Week 48
Population: mITT-E Population.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Scores on a scale
  Week 24, n=217, 213: number analyzed (Participants) | 217 | 213
  Week 24, n=217, 213 | 0.00 (0.012) | 0.02 (0.012)
  Week 48, n=224, 217: number analyzed (Participants) | 224 | 217
  Week 48, n=224, 217 | 0.01 (0.012) | 0.01 (0.012)

13. Secondary Outcome: Change From Baseline in EQ-5D Thermometer Scores at Week 24 and Week 48
Description: The European Quality of Life -5 Dimensions (EQ-5D) is a 5-question quality of life instrument that provides a utility score and visual analogue scale score that describes the participants' health status. The primary reason for including the EQ-5D is to elicit utility values for potential cost-effectiveness analysis for submission to health technology assessment agencies. Thermometer score is based on a visual analogue scale (VAS) ranging from 100 (best imaginable health state) to 0 (worst imaginable health state).Values represented are for adjusted mean. Estimates are calculated from an ANCOVA model adjusting for age, sex, race, Baseline viral load, background dual NRTI therapy and Baseline EQ-5D thermometer score. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Time Frame: Baseline, Week 24, and Week 48
Population: mITT-E Population.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 242 | 242
Scores on a scale
  Week 24, n=221, 216: number analyzed (Participants) | 221 | 216
  Week 24, n=221, 216 | 4.95 (0.885) | 5.96 (0.895)
  Week 48, n=224, 220: number analyzed (Participants) | 224 | 220
  Week 48, n=224, 220 | 5.78 (0.762) | 6.95 (0.769)

14. Secondary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Total Score at Week 4, Week 24, and Week 48
Description: Participant treatment satisfaction was measured using the self-reported scale (HIVTSQ), which consists of 10 items (1-satisfaction, 2-HIV control, 3-adverse effects, 4-level of demand, 5-convenience, 6-flexibility, 7-knowledge, 8-life habits, 9-recommendability, and 10-willingness to continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The treatment satisfaction score (range: 0-60) was the sum of the individual items. HIVTSQ mITT-E Population=Only participants from USA, France, Germany, Italy, Spain for whom valid translations were available from the mITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits, so the overall number of participants analyzed reflects everyone in the HIVTSQ mITT-E population.
Time Frame: Week 4, Week 24, and Week 48
Population: HIVTSQ mITT-E Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 214 | 206
Scores on a scale
  Week 4, n=206, 192: number analyzed (Participants) | 206 | 192
  Week 4, n=206, 192 | 54.1 (6.43) | 52.4 (7.94)
  Week 24, n= 211, 200: number analyzed (Participants) | 211 | 200
  Week 24, n= 211, 200 | 56.1 (5.16) | 54.3 (6.94)
  Week 48, n=212, 201: number analyzed (Participants) | 212 | 201
  Week 48, n=212, 201 | 56.1 (4.60) | 54.5 (6.78)

15. Secondary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Lifestyle/Ease Sub Score at Week 4, Week 24, and Week 48
Description: Participant treatment satisfaction was measured using the self-reported scale (HIVTSQ), which consists of 10 items (1-satisfaction, 2-HIV control, 3-adverse effects, 4-level of demand, 5-convenience, 6-flexibility, 7-knowledge, 8-life habits, 9-recommendability, and 10-willingness to continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The lifestyle/ease score is the sum of items 4, 5, 6, 7 and 8 (range: 0-30). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits, so the overall number of participants analyzed reflects everyone in the HIVTSQ mITT-E population.
Time Frame: Week 4, Week 24, and Week 48
Population: HIVTSQ mITT-E Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 214 | 206
Scores on a scale
  Week 4, n=202, 190: number analyzed (Participants) | 202 | 190
  Week 4, n=202, 190 | 26.7 (3.61) | 25.8 (4.48)
  Week 24, n=210, 199: number analyzed (Participants) | 210 | 199
  Week 24, n=210, 199 | 27.5 (3.16) | 26.6 (4.11)
  Week 48, n=211, 201: number analyzed (Participants) | 211 | 201
  Week 48, n=211, 201 | 27.6 (3.00) | 26.6 (4.11)

16. Secondary Outcome: Human Immunodeficiency Virus Treatment Satisfaction Questionnaire (HIVTSQ) Convenience Score at Week 4, Week 24, and Week 48
Description: Participant treatment satisfaction was measured using the self-reported scale (HIVTSQ), which consists of 10 items (1-satisfaction, 2-HIV control, 3-adverse effects, 4-level of demand, 5-convenience, 6-flexibility, 7-knowledge, 8-life habits, 9-recommendability, and 10-willingness to continue). Items are scored from 0 (very dissatisfied) to 6 (very satisfied), other than item 4, which has an inverted score from 6 (very demanding) to 0 (very undemanding). The convenience score is the score for item 5 (range: 0-6). Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed for different visits, so the overall number of participants analyzed reflects everyone in the HIVTSQ mITT-E population.
Time Frame: Week 4, Week 24, and Week 48
Population: HIVTSQ mITT-E Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DTG 50 mg QD | DRV 800 mg + RTV 100 mg QD
Number analyzed (Participants) | 214 | 206
Scores on a scale
  Week 4, n=204, 190: number analyzed (Participants) | 204 | 190
  Week 4, n=204, 190 | 5.6 (0.71) | 5.2 (1.11)
  Week 24, n=211, 200,: number analyzed (Participants) | 211 | 200
  Week 24, n=211, 200, | 5.6 (0.64) | 5.4 (1.01)
  Week 48, n=212, 201: number analyzed (Participants) | 212 | 201
  Week 48, n=212, 201 | 5.7 (0.62) | 5.4 (1.02)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) are presented from the available safety data from the start of the study medication up to end of study.
Description: SAEs and non-serious AEs were reported for members of the Modified Safety Population, comprised of all participants who received at least one dose of investigational product excluding one participant at one site, which was closed due to GCP non-compliance issues in another ViiV Healthcare sponsored trial.
Groups:
- DTG 50mg QD: Participants received DTG 50 mg QD administered in combination with FDC dual NRTI therapy (either ABC/3TC or TDF/FTC) for 96 weeks. Participants were then given the opportunity to receive DTG 50 mg QD during an Extension Phase of the study.
Arm/Group | DTG 50mg QD | DRV 800 mg + RTV 100 mg QD | Extension DTG 50 mg
All-Cause Mortality (participants affected / at risk) | 1/242 | 0/242 | 0/123
Serious Adverse Events (participants affected / at risk) | 36/242 | 21/242 | 4/123
Other Adverse Events (participants affected / at risk) | 221/242 | 214/242 | 52/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 50mg QD (N=242) | DRV 800 mg + RTV 100 mg QD (N=242) | Extension DTG 50 mg (N=123)
Suicide attempt (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Complication of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug use disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Proctitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG 50mg QD (N=242) | DRV 800 mg + RTV 100 mg QD (N=242) | Extension DTG 50 mg (N=123)
Diarrhoea (Gastrointestinal disorders) | 43 (46) | 74 (98) | 2 (2)
Nausea (Gastrointestinal disorders) | 40 (45) | 48 (56) | 2 (2)
Headache (Nervous system disorders) | 40 (45) | 26 (29) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 26 (33) | 24 (26) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 16 (22) | 27 (30) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 19 (21) | 1 (1)
Insomnia (Psychiatric disorders) | 19 (21) | 16 (17) | 1 (1)
Pyrexia (General disorders) | 16 (17) | 16 (17) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (16) | 17 (22) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 17 (17) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (19) | 0 (0)
Bronchitis (Infections and infestations) | 12 (12) | 17 (20) | 0 (0)
Fatigue (General disorders) | 15 (17) | 14 (15) | 0 (0)
Gastroenteritis (Infections and infestations) | 12 (13) | 14 (16) | 3 (3)
Dizziness (Nervous system disorders) | 14 (15) | 13 (14) | 0 (0)
Pharyngitis (Infections and infestations) | 11 (11) | 14 (15) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 12 (12) | 0 (0)
Syphilis (Infections and infestations) | 11 (12) | 12 (12) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 15 (19) | 0 (0)
Anxiety (Psychiatric disorders) | 13 (13) | 9 (9) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (10) | 13 (17) | 1 (1)
Sinusitis (Infections and infestations) | 9 (10) | 13 (14) | 0 (0)
Depression (Psychiatric disorders) | 12 (14) | 8 (9) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (13) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10) | 0 (0)
Asthenia (General disorders) | 5 (7) | 11 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (13) | 5 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (12) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 8 (10) | 9 (9) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 10 (10) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 11 (11) | 2 (2)
Flatulence (Gastrointestinal disorders) | 5 (6) | 11 (11) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 8 (8) | 6 (6) | 1 (1)
Influenza like illness (General disorders) | 9 (11) | 6 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 4 (4) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 8 (9) | 0 (0)
Folliculitis (Infections and infestations) | 7 (7) | 6 (6) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 0 (0)
Urethritis (Infections and infestations) | 8 (8) | 4 (4) | 1 (1)
Conjunctivitis (Infections and infestations) | 4 (4) | 7 (7) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 8 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 7 (9) | 0 (0)
Gonorrhoea (Infections and infestations) | 8 (9) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (9) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 9 (9) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 6 (6) | 1 (1)
Rhinitis (Infections and infestations) | 4 (4) | 6 (8) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (5) | 0 (0)
Chest pain (General disorders) | 3 (3) | 7 (8) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (8) | 4 (4) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 5 (5) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 6 (7) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) | 1 (1)
Tonsillitis (Infections and infestations) | 5 (5) | 3 (4) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 4 (5) | 4 (4) | 0 (0)
Oral herpes (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Pain (General disorders) | 3 (3) | 5 (6) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (3) | 5 (5) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4) | 0 (0)
Furuncle (Infections and infestations) | 3 (3) | 4 (5) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Seasonal allergy (Immune system disorders) | 3 (3) | 3 (3) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 5 (7) | 1 (1)
Viral infection (Infections and infestations) | 6 (6) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0)
Acarodermatitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 0 (0)
Chills (General disorders) | 2 (2) | 4 (4) | 0 (0)
Chlamydial infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Drug use disorder (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 4 (5) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 4 (5) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 0 (0)
Hypersensitivity (Immune system disorders) | 4 (5) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 4 (4) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0)
Malaise (General disorders) | 3 (3) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 2 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (5) | 0 (0)
Peripheral swelling (General disorders) | 3 (3) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Weight increased (Investigations) | 3 (3) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (3) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Genital herpes (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 0 (0)
Herpes simplex (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1)
Hypogonadism (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0)
Multiple allergies (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Sleep disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Body tinea (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatophytosis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 2 (3) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Local swelling (General disorders) | 1 (1) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 1 (4) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (3) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (4) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Burn oral cavity (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ear infection fungal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Latent tuberculosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Libido disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Renal tubular dysfunction (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0)
Secondary syphilis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Tobacco abuse (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess sterile (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Asthenospermia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bereavement (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Burnout syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Campylobacter test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Condyloma latum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysplasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ear canal erythema (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Ejaculation failure (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection syphilitic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Family stress (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flat affect (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Latent syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lipids increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymph node palpable (Investigations) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucocutaneous ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oropharyngitis fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Parasite stool test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Penis injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pityriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Primary syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Product use complaint (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rectal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Scleral discolouration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sports injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Strongyloidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Submandibular mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Substance use (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Substance use disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tic (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar exudate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Ureaplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.